CLINICAL TRIAL: NCT03015935
Title: Safe and Easy Access Technique for the First Trocar in Laparoscopic Obesity Surgery. A Prospective Controlled-cohort Study
Brief Title: Safe and Easy Access Technique for the First Trocar in Laparoscopic Obesity Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Fatih Basak, Medical Doctor, Umraniye Education and Research Hospital
Other Study IDs: First_Trocar_Entery
Record Dates: First submitted 2017-01-03; First posted 2017-01-10 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Obesity, Morbid
Keywords: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Optical: visual-assisted entry
  Interventions: Procedure: visual-assisted entry
- Veress: Veress entry
  Interventions: Procedure: Veress entry

INTERVENTIONS:
Procedure: visual-assisted entry — First trocar entry will be performed with visual-assisted trocar
  Groups: Optical
Procedure: Veress entry — First trocar entry will be performed with Veress
  Groups: Veress

SUMMARY:
Laparoscopic surgery has become very popular and standard in many indications after advancements of technique. Various methods have been used in first entry to the abdomen. Safety, wound size, to be not time-consuming, low cost, learning curve and efficacy are important. Several techniques, instruments, and approaches to minimize the risk of injury (the bowel, bladder, major abdominal vessels, and an anterior abdominal wall vessel) have been introduced.

There is no consensus yet on an optimal method has yet emerged.

The investigators aimed to evaluate efficacy of entry methods that ensures safe insertion of the first trocar at any site of the abdomen.

To evaluate the efficacy of entry technique, the investigators used cohort of patients who will be planned to laparoscopic obesity surgery.

Two methods are commonly used in surgical literature and in our center.

The investigators have been used visible optical-entry technique in some patients for first entry and Veress technique in some other patients.

For this purpose, the investigators designed an observational study.

DETAILED DESCRIPTION:
Several techniques, instruments, and approaches to minimize the risk of injury (the bowel, bladder, major abdominal vessels, and an anterior abdominal wall vessel) have been introduced.

These methods include the standard technique of insufflation after insertion of the Veress needle, the open (Hasson technique), the direct trocar insertion and optical trocar insertion. Furthermore, it is more difficult to perform in the obese patient, especially if the first trocar is not umbilical, like obesity surgery. This is because obese patients have a very thick abdominal wall (particularly in women) as well as a thick peritoneum.

Very different complications, some even potentially fatal, i.e., injury to viscera or to major intra-abdominal and abdominal wall vessels, have been reported in surgical literature. Complications of first entry develop in up to 1-2% of patients and more than half of all are fatal complications. Major vascular and abdominal organ injury rates of 0.03-0.1% and 0.08-0.14%, respectively, have been reported. Surprisingly, there has been little change in entry techniques since the dawn of laparoscopic surgery. Some risk factors are defined for prediction of complications, such as obesity. Laparoscopic obesity surgery has become very attractive and gaining popularity, recently, and however it possess many complications and challenges such as (it starts with) entry to the abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with body mass index of >40

Exclusion Criteria:

* Patients who have skin disease at operation area

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are eligible for laparoscopic obesity surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Entry time | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Basak, Study Chair — Umraniye Education and Research Hospital
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No